CLINICAL TRIAL: NCT02738021
Title: Stepped Care for Postpartum Depression in Pediatric Primary Care: A Pilot Project at Gouverneur Health Services
Brief Title: Managing PPD at Gouverneur
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00416
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Post-Partum Depression
Keywords: Psychosocial; Psychotherapy; Maternal
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STRONG (Experimental): A brief 3-session IPT-based preventive intervention, on maternal and child health outcomes.
  Interventions: Behavioral: STRONG

INTERVENTIONS:
Behavioral: STRONG — A brief 3-session IPT-based preventive intervention, on maternal and child health outcomes.

SUMMARY:
A Stepped Care pathway for managing postpartum depression (PPD) in pediatric primary care settings will be used to (1) understand context for implementation feasibility (2) evaluate benefits for mother and child.

The proposed pilot project will be conducted as part of a quality improvement effort in the Department of Pediatrics at Gouverneur Health Services to improve management of postpartum depression during pediatric primary care visits. This project will test the feasibility of a stepped care approach to identifying and managing depression among mothers of infants (0-6 months). This study will provide preliminary data on the feasibility of the care management protocol, implementation and fidelity measures, and training/consultation methods within a real world pediatric care practice. These data will inform and support the preparation of a large-scale NIH grant.

Specific research questions include:

1. To pilot the feasibility of using a Stepped Care Approach to identify and mange maternal depression within primary care pediatric care visits, with a focus on mothers of infants 0-6 months.

   1. Train non specialty MH providers to systematically identify maternal depression.
   2. Assess how effective integration of maternal depression intervention is as part of well baby visits.
2. To o examine the impact of STRONG, a brief 3-session IPT-based preventive intervention, on maternal and child health outcomes (e.g., maternal depression symptoms, child receipt of acute care services). Secondary outcomes include maternal social support and parenting practices.

ELIGIBILITY:
Inclusion Criteria for Subjects

* PHQ-9 scores in the 10-19 range
* Women with infants 6 months and younger at time of screening

Inclusion Criteria for Providers

Exclusion Criteria:

* Active substance use
* Current treatment for depression
* Current/past history of schizophrenia, bipolar or other psychotic disorder;
* Suicidal/Homicidal risks;
* Women with difficulties speaking or understanding English;
* Women under the age of 18.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | One year
  A validated 9-item self-administered version of the PRIME-MD that assesses depression severity.

SECONDARY OUTCOMES:
Maternal Depression Management Inventory | One year
  It is a fifty-nine (59) item survey of primary care provider beliefs, attitudes and practices related to the assessment and management of maternal depression.

CONTACTS AND LOCATIONS:
Overall Officials: Serene Olin, PhD, Principal Investigator — NYU Langone Health